CLINICAL TRIAL: NCT06390553
Title: Effect of Task-Oriented Virtual Reality Access With Crowd Simulation on Freezing Phenomenon, Balance, Functional Mobility, Participation and Quality of Life in Parkinson's Patients
Brief Title: Effect of Virtual Reality on Freezing Phenomenon, Balance, Functional Mobility, Participation in Parkinson's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ertuğrul Demirdel, Assoc. Prof., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraYBÜ-VR
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease; Freezing of Gait
Keywords: virtual reality; rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): Patients in the conventional treatment group will be given 15 minutes of walking training in addition to the 45 minutes of conventional Parkinson's rehabilitation program. Patients in the conventional treatment group will be trained in flexibility (lumbar extensors, hip flexors, hamstrings, pectorals), balance (weight transfer, static balance with stress loading) coordination (rotational and bilateral activities), respiratory (thoracic expansion, respiratory control), strength (hip circumference, abdomen, back extensors), stabilization, posture (chin tuck, scapular adduction) exercises will be given and the number of repetitions will be adjusted according to patient performance.
  Walking training to be given to the conventional group will include walking in different directions, walking with arm swing, walking over blocks, stopping and restarting walking, and changing direction activities.
  Interventions: Procedure: Conventional Parkinson Rehabilitation
- Virtual reality group (Experimental): Patients in the virtual reality group will be given a 45-minute conventional Parkinson's rehabilitation program similar to those in the conventional group, followed by 15 minutes of virtual reality walking training. Patients in the virtual reality group will be trained in flexibility (lumbar extensors, hip flexors, hamstrings, pectorals), balance (weight transfer, static balance with stress loading) coordination (rotational and bilateral activities), Respiratory (thoracic expansion, respiratory control), strength (hip circumference, abdomen, back extensors) stabilization, posture (chin tuck, scapular adduction) exercises will be given and the number of repetitions will be adjusted according to patient performance. Virtual reality applications increase the sense of reality in the individual with enriched virtual environments where sensory inputs are increased and provide the opportunity to perform activity training with a rich variety of tasks.
  Interventions: Device: Task-Oriented Virtual Reality Application with Crowd Simulation; Procedure: Conventional Parkinson Rehabilitation

INTERVENTIONS:
Device: Task-Oriented Virtual Reality Application with Crowd Simulation — Patients will be treated 4 days a week for 8 weeks in accordance with their assigned group.
  Arms: Virtual reality group
Procedure: Conventional Parkinson Rehabilitation — Patients will be treated 4 days a week for 8 weeks in accordance with their assigned group.

SUMMARY:
This study was planned to investigate the use and results of virtual reality applications with specially prepared software for the rehabilitation of freezing phenomenon, which increases the falling anxiety of individuals with Parkinson's disease and causes social isolation. Individuals over the age of 50 who have been diagnosed with idiopathic Parkinson's disease by a specialist neurologist will be included in the study; Individuals evaluated in terms of balance, functional mobility, freezing phenomenon, participation, and cognitive status will be randomly divided into two groups receiving conventional treatment and additional virtual reality. After the preliminary evaluation, they will receive 8 weeks of treatment 4 days a week and will be evaluated after the treatment and 3 months after the treatment. In addition to the improvements that will emerge as a result of the treatments within the scope of the study, it is expected that the virtual reality application created with crowd simulation will provide more effective results in improving the parameters. Knowing the effects of exercises in crowds, which cannot be performed in the clinic, in the treatment of Parkinson's disease patients, whose freezing and freezing-related symptoms are aggravated, especially in crowded environments, will make significant contributions to the field.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Parkinson's disease by a qualified neurologist (diagnosed with idiopathic PD according to UK Brain Bank criteria
* Being between 1-2.5 stages according to the Hoehn and Yahr Staging Scale
* Volunteering to participate in the study
* 50 years of age or older
* Standardized Mini Mental Test score greater than 24
* Patients experiencing an on-off period are in the "on" period
* Not using deep brain stimulation or drug pump
* Ability to walk independently on level ground (Functional Ambulation 3 and above according to classification)
* Having a score of (≥2) on item 3 of the freezing while walking scale

Exclusion Criteria:

* Being any neurological or psychiatric disease other than Parkinson's disease
* Cardiovascular, vestibular or musculoskeletal disease
* Dyskinetic movements
* Having vision problems that cannot be corrected with glasses or lenses
* Hearing problems that cannot be corrected with a hearing aid
* Using an assistive device

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Freezing Phenomenon | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  The presence and severity of freezing in patients will be evaluated with the Freezing of Gait Questionnaire. It consists of six items and each item is evaluated with a 5-point Likert scale. In the scale, which was adapted into Turkish by Candan et al., the score range is 0-24 and high scores indicate that the condition associated with frostbite is poor.
Balance | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  The balance of the patients will be evaluated with the Biodex Balance System. Postural stability and fall risk will be evaluated.
Functional Mobility | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  The Timed Get Up and Go Test (TUG) will be used to assess functional mobility. The TUG, which includes walking and turning functions, has been shown to be highly reliable and valid for individuals with Parkinson's disease). The person to be tested sits on a chair at normal height. With the command "Go", the person is asked to get up from the chair and walk 3 m forward at a normal walking speed and then return and sit back on the chair. It is usually administered twice and the average time is recorded. The person is allowed to use an assistive device (if available) and this is noted.
Quality of Life Assessment | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  Quality of life will be assessed with Parkinson's Disease Questionnaire (PDQ-8) developed specifically for individuals with Parkinson's disease. This validated questionnaire consists of eight questions to assess mobility, activities of daily living, emotional well-being, disease stigma, social support, cognition, communication and physical discomfort . In the questionnaire, the status of the person in the last month is questioned. The total score is between 0 and 100, with lower scores indicating better perceived health status due to the disease.
Participation | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  In order to evaluate social participation in the study, home participation (grocery shopping, meal preparation, daily household chores, money management, etc.), social participation (hobby, going out of the house, etc.), productivity (school, work, volunteer activities, etc.), electronic A scale consisting of 43 social networks (internet use, social communication, mobile phone use, etc.), 4 subunits and a total of 18 questions will be used.

SECONDARY OUTCOMES:
Executive functions | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  The Trail Making Test (TMT) will be used to assess executive functions. The TMT measures executive functions such as working memory, complex attention, planning and set switching and requires visual-spatial processing and motor skills. TMT , A and B It consists of two parts. Part A of the TMT, which is an executive function test, evaluates the processing speed based on visual scanning ability, while part B evaluates the ability to change the setup between stimulus sets and to follow the sequentiality. Cangöz et al. determined the standardized values of the test for people over 50 years of age.
The activity-specific balance confidence scale | Day 1-Study Day Visit; 8-week Follow-up Visit; 3-month Follow-up Visit
  The activity-specific balance confidence scale will be used to assess the level of confidence the individual feels when performing balance-related activities of daily living. In the questionnaire consisting of 16 questions, the level of confidence felt ranges from 0% (completely insecure) to 100% (completely safe). The score obtained is divided by 16 to obtain a total score. 0-49 points indicate low functional level, 50-80 points indicate medium functional level and 81-100 points indicate high functional level. Scores below 67% indicate a fall risk in elderly individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul DEMİRDEL, Assoc. Prof., Study Director — Ankara Yildirim Beyazıt University; Özge BARUT ÇELİK, MSc., Study Chair — Kirsehir Ahi Evran University; Figen TUNCAY, Prof., Principal Investigator — Kirsehir Ahi Evran University; Öner BARUT, Asst. Prof., Principal Investigator — Gazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Gazi University, Ankara, Maltepe
  - Kirsehir Ahi Evran University, Kirşehi̇r, Merkez
  - Ankara Yildirim Beyazit University, Ankara, Çubuk